CLINICAL TRIAL: NCT06901206
Title: Neonatologist-Performed Lung Ultrasound (NPLUS) to Guide Respiratory Therapy on Non-Invasive Ventilation in Preterm Infants
Brief Title: Neonatologist-Performed Lung Ultrasound (NPLUS) to Guide Respiratory Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Hospital For Women (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Tim Schindler, Senior Staff Specialist, Royal Hospital for Women; Conjoint Associate Professor, University of New South Wales, Royal Hospital For Women
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024/PID01756
Record Dates: First submitted 2025-03-10; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: PreTerm Neonate; Respiratory Distress Syndrome (RDS)
Keywords: NPLUS; Neonatologist performed lung ultrasound; lung ultrasound score; CPAP; loss of aeration; atelectasis; preterm neonate; respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome; Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NPLUS (Active Comparator): In the NPLUS block, lung ultrasound is performed at T0 (reported persistent increased FiO2 demand) and T1 (one hour after T0). NPLUS may be able to detect loss of aeration and lead to more targeted interventions to improve lung aeration.
  Interventions: Procedure: Neonatologist performed lung ultrasound
- Control (No Intervention): Routine Care

INTERVENTIONS:
Procedure: Neonatologist performed lung ultrasound — Neonatologist performed lung ultrasound is performed at T0 (reported persistent increased FiO2 demand) and T1 (one hour after T0). NPLUS may be able to detect loss of aeration and lead to more targeted interventions to improve lung aeration. A comprehensive lung ultrasound examination will take 5 minutes or less to perform and involves minimal handling for the patient.
  Arms: NPLUS

SUMMARY:
The goal of this cross-over clinical trial is to evaluate whether Neonatologist-Performed Lung Ultrasound (NPLUS) can be used in preterm babies on non-invasive breathing support to reduce the amount of oxygen they need. The main question it aims to answer is:

When a baby's oxygen requirement goes up, does NPLUS help to target interventions and reduce oxygen requirements?

Researchers will compare NPLUS to standard treatment.

Participants will:

Have a lung ultrasound performed whenever their oxygen requirement increases by more than 10%.

The ultrasound findings will be used to target interventions that aim to improve air entry in the lungs.

Each time this happens, the researchers will note what happens to the oxygen requirement afterwards.

Each participant will participate for five days. For the first two days, they will be randomized to either the NPLUS arm or the usual care arm.

There is then a 24 hour period of usual care. For the final two days, participants cross over to the other arm of the trial.

DETAILED DESCRIPTION:
NPLUS is used to detect various artifacts that emerge due to air and fluid ratio in the lungs. The image results form a beam reflection and reverberation of echoes on tissues. The most important artifacts display A-lines, B-lines and the pleural line with the lung sliding. A-lines (horizontal, hyperechogenic long line reverberation artefacts of the pleura) are a sign of aeration. B-lines (vertical, hyperechoic ring-down artefacts arising from the pleural line) indicate fluid in the interstitial space. The pleural line is a smooth, hyperechoic line. Breathing or ventilation causes a movement of the pleural sheets resulting in a visible sliding as definitive sign of lung aeration and ventilation.

Lung consolidations can be sonographically detected by an absence of the pleural line and therefore the lung sliding and areas with loss of aeration visible as lung with tissue like density. Consolidations can be caused by several conditions (e.g., atelectasis, pneumonia, contusion) and the differentiation can be done by ultrasound.

Preterms are prone for recurrent episodes of loss of aeration due to small airway size and muscular weakness. Lung ultrasound has established in the last years and has become an emerging tool for bedside evaluation and to dynamically assess the lungs in several respiratory conditions. Detecting loss of aeration via lung ultrasound is fast and feasible. Trials have investigated the role of lung ultrasound to guide surfactant admission and extubation failure.

To our knowledge there is no evidence investigating the feasibility of lung ultrasound to guide respiratory therapy for preterms on non-invasive ventilation. Oxygen exposure is associated with numerous complications in preterms and should be maintained as low as possible. Lung ultrasound could be a promising tool for a faster detection of loss of aeration and due to more targeted intervention with the ultrasound knowledge a faster FiO2 reduction could be achieved.

The main objective of this study is to evaluate, if NPLUS performed according to a standardized protocol (lung ultrasound score, LUS) in preterm neonates with an absolute increase ≥ 10% over their baseline FiO2 on non-invasive ventilation can detect loss of aeration resulting in more effective reduction of FiO2 demand through targeted interventions (e.g., temporary PEEP increase for alveolar recruitment, positioning of the patient) compared to routine care.

The present study is a cross-over study evaluating the use of NPLUS to guide respiratory therapy of preterm infants on non-invasive ventilation. After inclusion of the study patient, an observation time of two 48-hour blocks and a washout phase of 24 hours between these two blocks is set. Each 48-hour block is managed according to the assigned treatment (NPLUS or standard care). In the 24-hour washout phase no study-related interventions are performed. The treatment assignments are swapped after the washout phase and in the next 48 hours infants previously assigned to NPLUS receive standard care and infants previously assigned to standard care receive NPLUS. Within these set time periods, each episode of increased persisting (>10 min) FiO2 demand (absolute increase ≥ 10% over the FiO2 baseline) on non-invasive ventilation is defined as event (e.g., patient 1, event 1). For each event, T0 is the time point when the absolute increase ≥ 10% over the initial FiO2 baseline was reported to the clinician and an intervention may be initiated, and T1 is the time point 1 h after T0. The clinician in charge is informed about the onset of every single event. In both treatment arms, interventions for every occurring event can be considered by the clinician in charge including targeted repositioning of the patient, temporary PEEP increase for alveolar recruitment, changes in ventilatory settings (e.g. change to Bilevel, NIPPV, NAVA), surfactant therapy, indication for a chest x-ray, and indication for thoracic physiotherapy.) In the 48-hour NPLUS block, lung ultrasound is performed at T0 (reported persistent increased FiO2 demand) and T1 (one hour after T0). NPLUS may be able to detect loss of aeration and lead to more targeted interventions to improve lung aeration. A comprehensive lung ultrasound examination will take 5 minutes or less to perform and involves minimal handling for the patient.

For each subject a baseline FiO2 is established for the control and NPLUS periods. The aim of using NPLUS versus standard care when managing an event is to reduce any increase from the subject's baseline in the resolution FiO2 level associated with the event.

The ratio of the FiO2 at resolution of each event to baseline FiO2 is a continuous measurement which is 1 when the resolution FiO2 equals the subject's baseline value. A ratio of 1.2 means the resolution FiO2 for the event is 20% higher than the subject's baseline FiO2, a ratio <1 indicates the resolution FiO2 for the event is less than the subject's baseline and so on.

ELIGIBILITY:
Inclusion Criteria:

* All preterm infants (<33 weeks gestational age) from their 2nd week of life, receiving respiratory support via NCPAP
* expected to stay on NCPAP for the following 5 days at the NICU, Royal Hospital for Women, Randwick, Sydney
* provided written informed consent obtained from parents.

Exclusion Criteria:

* Neonates with previous abdominal surgery
* Major congenital anomalies.
* >33+0 weeks
* Less than 1 week of age
* Invasive ventilation
* Bilevel or Multilevel non-invasive ventilation
* Not expected respiratory support via CPAP for the following 5 days.

Min Age: 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mean ratio res/base (Resolution FiO2 / Baseline FiO2) | Resolution FiO2 assessed 1 hour after increased persisting (>10 min) FiO2 demand (absolute increase ≥ 10% over the FiO2 baseline)
  For each subject a baseline FiO2 is established for the control and NPLUS periods. Each episode of increased persisting (>10 min) FiO2 demand (absolute increase ≥ 10% over the FiO2 baseline) on non-invasive ventilation is defined as event.
  The aim of using NPLUS versus standard care (control) when managing an event is to reduce any increase from the subject's baseline in the resolution FiO2 level associated with the event.
  The ratio of the FiO2 at resolution of each event to baseline FiO2 is a continuous measurement which is 1 when the resolution FiO2 equals the subject's baseline value. A ratio of 1.2 means the resolution FiO2 for the event is 20% higher than the subject's baseline FiO2, a ratio <1 indicates the resolution FiO2 for the event is less than the subject's baseline and so on.

SECONDARY OUTCOMES:
Mean FiO2 (within 48-hour blocks) | 48 hours
  comparison of infants mean FiO2 in NPLUS vs. control period
FiO2 between T0 and T1 | Assessed 1 hour after increased persisting (>10 minutes) FiO2 demand (absolute increase ≥ 10% over the FiO2 baseline)
LUS between T0 and T1 | Assessed 1 hour after increased persisting (>10 minutes) FiO2 demand (absolute increase ≥ 10% over the FiO2 baseline)
Number of changes in ventilatory settings (PEEP) | 48 hours
  Total number of changes from baseline PEEP settings during each study period.
SpO2/FiO2 ratio | 48 hours
Routinely obtained capillary blood gas analysis (pH, pCO2) | 48 hours
  at certain time points within the study period.
Number of chest X-rays and NPLUS examinations, number of chest X-ray based interventions, number of NPLUS based interventions. | 48 hours
Number of recruitment maneuvers | 48 hours
  Number of recruitment maneuvers (e.g., repositioning of the patient, temporary PEEP increase for alveolar recruitment, changes in ventilatory settings (e.g.change to Nava), surfactant therapy, indication of a chest x-ray, and indication of thorax physiotherapy).
Time to detect impairment of lung aeration (consolidations). | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tim Schindler BMedSc MBBS FRACP PhD, Principal Investigator — Senior Staff Specialist, Royal Hospital for Women, Conjoint Associate Professor, University of New South Wales
Locations (1):
- Newborn Intensive Care Unit, Royal Hospital for Women, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No